CLINICAL TRIAL: NCT02628275
Title: Will Mild vs. Moderate Physical Activity Suffice to Abate the Progression of Subclinical Atherosclerosis in Sedentary Adults?
Brief Title: Impact of Mild or Moderate Physical Activity and Progression of Subclinical Atherosclerosis
Acronym: MoMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Eric Larose, DVM, MD, FRCPC, FCCS, FAHA, Full Professor, Faculty of Medicine, Laval University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CIHR MOP-137079
Record Dates: First submitted 2015-11-26; First posted 2015-12-11 (Estimated); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Atherosclerosis
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention): Continued inactivity
- Moderate to vigorous physical activity (Active Comparator): MVPA (55-90% of maximum heart rate) for 150 min/week (current recommendations)
  Interventions: Behavioral: Moderate to vigorous physical activity
- Light physical activity (Active Comparator): LPA (40-55% of maximum heart rate) for 150 min/week
  Interventions: Behavioral: Light physical activity

INTERVENTIONS:
Behavioral: Moderate to vigorous physical activity — 55-90% maximum heart rate for 150min/week (current recommendations)
  Arms: Moderate to vigorous physical activity
Behavioral: Light physical activity — 40-55% maximum heart rate for 150min/week
  Arms: Light physical activity

SUMMARY:
Subclinical atherosclerosis is identified in roughly 2/3rd of otherwise healthy young adults. How much physical activity is required to prevent progression of subclinical atherosclerosis? In the 85% of healthy younger Canadian men and women who do NOT perform the recommended 150 min/week of moderate- to vigorous-intensity physical activity (MVPA) as recommended, is it reasonable to aim for a lower regimen of light physical activity (LPA) despite the absence of supporting literature, or to the contrary should the investigators insist on achieving MVPA? In this perspective, MoMA provides a unique opportunity to determine whether LPA vs. MVPA is necessary to limit subclinical atherosclerosis progression in inactive otherwise healthy adults. Resolving such unknowns should inform strategies to prevent decades of silent disease progression leading to future morbidity and mortality.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) remains rampant in developed regions, topping the list of causes of mortality leading to 29% of all deaths. In addition to mortality, the economic impact of morbidity and hospitalization related to CVD costs Canadians over $22.2 billion every year. By far the leading cause of CVD is atherosclerosis defined as a thickening of the arterial wall with fatty deposits. Therefore, atherosclerosis is the underlying mechanism behind the #1 cause of mortality and morbidity in developed regions. Autopsy studies performed in healthy casualties of the Korean, Vietnam, Iraq and Afghanistan Wars revealed that atherosclerosis is present in up to 78% of young men before their 30th birthday, even in the absence of traditional risk factors (high blood pressure, dyslipidemia, obesity). Prevention of atherosclerosis and its silent progression towards clinical events decades later should therefore become a priority in all young adults. A potentially powerful avenue of cardiovascular prevention lies in the reduction of subclinical atherosclerosis progression in younger adults through physical activity. Unfortunately, only 15% of Canadians meet the current recommendations for 150min/week of moderate- to vigorous-intensity physical activity (MVPA). In response to the observation that Canadians simply don't find time for/or do not appear to value current recommendations, it was suggested that even light-intensity physical activity (LPA) might improve biomarker levels compared to a sedentary lifestyle. It appears that in the face of failed attempts to convince Canadians to perform 150min/week of MVPA, expectations towards LPA have been lowered despite the absence of convincing data.

MoMA is a randomized controlled trial to study the effects of two doses of physical activity on subclinical atherosclerosis burden progression; 270 inactive men and women aged 18-40 years without CVD or risk factors will be enrolled. At baseline, risk factors, physical activity level and nutritional habits will be measured through validated questionnaires; blood work and anthropometric parameters measurements will be performed (markers of cardiometabolic risk); fitness level will be assessed through treadmill test and accelerometer; magnetic resonance imaging of carotid atherosclerosis, liver and adipose tissue will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Inactivity during leisure time as assessed through the long version of the International Physical Activity Questionnaire;
* Apparent health defined as 1) no known CVD (coronary, cerebrovascular or peripheral vascular disease), and 2) no known cardiovascular risk factors or cardiovascular medications (hypertension, dyslipidemia, diabetes, active smoking within past year, or clinical obesity defined as body mass index (BMI) ≥ 30kg/m2);
* Signed consent form.

Exclusion Criteria:

* Known dyslipidemia (participants receiving lipid-lowering medication, or in the absence of such medication, having: a fasting total plasma cholesterol level > 6.2 mmol/L, a triglyceride level ≥ 1.7 mmol/L, and/or HDL-cholesterol level < 1.0 mmol/L in men and < 1.3 mmol/L in women);
* Hypertension (participants receiving antihypertensive medications or having blood pressure ≥ 135/85 mmHg);
* Diabetes (participants taking diabetes medication or having plasma HbA1c ≥ 6.5%);
* Postmenopausal women;
* Pregnancy or nursing in the past year or expected in the next two years;
* Contraindications to MRI, as per the standardized IUCPQ MRI screening form;
* Participation in another research study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 129 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2022-10 (Actual); Study Completion 2022-10 (Actual)

PRIMARY OUTCOMES:
Change in carotid vessel wall volume measured by magnetic resonance imaging (MRI) | Baseline, 1 year, 2 years

SECONDARY OUTCOMES:
Change in waist circumference | Baseline, 1 year, 2 years
Change in hip circumference | Baseline, 1 year, 2 years
Change in BMI | Baseline, 1 year, 2 years
Change in abdominal visceral adipose tissue | Baseline, 1 year, 2 years
Change in abdominal subcutaneous adipose tissue | Baseline, 1 year, 2 years
Change in thoracic visceral adipose tissue | Baseline, 1 year, 2 years
Change in hepatic fat fraction | Baseline, 1 year, 2 years
Change in blood pressure | Baseline, 1 year, 2 years
Change in standard plasma lipid fractions | Baseline, 1 year, 2 years
Change in plasma apolipoprotein A1 | Baseline, 1 year, 2 years
Change in plasma apolipoprotein B | Baseline, 1 year, 2 years
Change in plasma lipid particle size | Baseline, 1 year, 2 years
Change in blood glucose | Baseline, 1 year, 2 years
Change in blood insulin | Baseline, 1 year, 2 years
Change in blood HbA1c | Baseline, 1 year, 2 years
Change in adiponectin | Baseline, 1 year, 2 years
Change in IL-6 | Baseline, 1 year, 2 years
Change in TNF-alpha | Baseline, 1 year, 2 years
Change in CRP | Baseline, 1 year, 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Eric Larose, DVM, MD, Principal Investigator — Institut universitaire de cardiologie et de pneumologie de Québec, University Laval
Locations (1):
- Institut universitaire de cardiologie et de pneumologie de Québec - Université Laval, Québec, Canada